CLINICAL TRIAL: NCT06933472
Title: A Randomized, Double-Blind, Multi-Regional, Phase 3 Study to Evaluate the Efficacy and Safety of AP301 on Serum Phosphorus Control in Chronic Kidney Disease Patients Receiving Maintenance Dialysis With Hyperphosphatemia
Brief Title: A Study of a Novel Iron-based Phosphate Binder AP301 in Patients With Hyperphosphatemia in the U.S. and China
Acronym: RESPOND-2
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alebund Pharmaceuticals (Industry)
Collaborators: Fortrea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AP301-HP-03
Record Dates: First submitted 2025-03-19; First posted 2025-04-18 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-06

CONDITIONS: Hyperphosphatemia; Chronic Kidney Disease, Receiving Dialysis; ESRD (End-Stage Renal Disease); Dialysis
Keywords: Hyperphosphatemia; AP301; Dialysis; ESKD
MeSH Terms: conditions — Hyperphosphatemia; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AP301 (Experimental): A blood phosphate-lowering medication containing iron
  Interventions: Drug: AP301
- AP301 Low Dose (Experimental): A blood phosphate-lowering medication containing iron, but with a low dose considered as ineffective
  Interventions: Drug: AP301 Low Dose

INTERVENTIONS:
Drug: AP301 — Three times a day, administered orally with three meals at a daily dose level from 2.7g to 9.0g
  Arms: AP301
Drug: AP301 Low Dose — Three times a day, administered orally with three meals at a daily dose level from 0.075g to 0.25g
  Arms: AP301 Low Dose

SUMMARY:
The goal of this clinical trial is to learn if AP301 could work in the patients receiving maintenance dialysis with elevated blood phosphate. The main questions it aims to answer are:

* Does AP301 lower blood phosphate levels?
* Does AP301 works on serum calcium level, calcium times phosphate level, and intact parathyroid hormone level?
* What discomfort or medical problem do the patients have when taking AP301?
* Does AP301 improve quality of life in Chinese patients?

The researchers will compare AP301 to an ineffective comparator (a look-alike substance that contains low dose AP301) to see if AP301 works to treat elevated blood phosphate.

In the study, the patients will experience the following stages in a chronicle order:

* Stop all using blood phosphate-lowering drugs,
* Take AP301 or the comparator three times a day for 8 weeks,
* Take AP301 three times a day for 24 weeks, and
* Take AP301 or the comparator three times a day for 3 weeks.

In the first 32 weeks, the dose of AP301 will be adjusted upwards or downwards based on the patient's blood phosphate level and the study doctor's judgment.

If the participant has a blood phosphate level above or below a certain level, they may receive additional treatment to lower the blood phosphate level.

ELIGIBILITY:
Key Inclusion Criteria:

* Provision of signed and dated ICF
* Age ≥ 12 years when signing the ICF
* Patients on dialysis for ≥ 3 months before signing the ICF and throughout the study
* For HD patients, spKt/V ≥ 1.2; for PD patients, total Kt/V ≥ 1.7/week
* Patients who receive phosphate-lowering drugs over 4 weeks and their serum phosphate level is:

  1. Screening: 1.13 mmol/L (3.5 mg/dL) ≤ serum phosphate < 2.58 mmol/L (8.0 mg/dL)
  2. After washout: 1.94 mmol/L (6.0 mg/dL) ≤ serum phosphate < 3.23 mmol/L (10.0 mg/dL)

Key Exclusion Criteria:

* History or plan of kidney transplantation
* History or plan of parathyroid intervention 6 months before signing the ICF
* Serum calcium < 1.9 mmol/L (7.6 mg/dL) or > 2.75 mmol/L (11 mg/dL) at screening
* Serum intact parathyroid hormone > 127 pmol/L (1200 pg/mL) at screening
* Presence of clinically significant gastrointestinal (GI) disorder
* History of gastrectomy or duodenectomy, or GI surgery within 3 months before signing the ICF
* Known allergic to any ingredient of AP301, or known history of severe allergies leading to emergency medical care
* Female who are breastfeeding

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 264 (Estimated)
Dates: Start 2025-06-13 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2027-01-10 (Estimated)

PRIMARY OUTCOMES:
Change in serum phosphate concentrations in the AP301 and the AP301 low dose groups | From Baseline to the end of Week 8
  The amount of phosphate in the blood will be measured with a standard laboratory test. The change in phosphate levels will be compared between the group receiving AP301 and the group receiving AP301 low dose.

SECONDARY OUTCOMES:
Chang in serum phosphate concentrations in the AP301 maintenance dose and the AP301 low dose groups | From the beginning of Week 33 to the end of Week 35
  The amount of phosphate in the blood will be measured with a standard laboratory test. The change in phosphate levels will be compared between the group receiving AP301 maintenance dose and the group receiving AP301 low dose.
Change in serum phosphate concentrations over time throughout the study | From Baseline to the end of Week 35
Change in serum calcium (Ca) and intact parathyroid hormone levels over time | From Baseline to the end of Week 35
  The amount of calcium and intact parathyroid hormone (iPTH) in the blood will be measured with standard laboratory tests.
Number of adverse events | From Baseline to Follow-up (Up to 37 weeks)
Change in QT intervals measured by 12-lead electrocardiagram test over time | From Baseline to the end of Week 35
  The duration of QT intervals will be measured with a standard 12-lead electrocardiagram test.

OTHER OUTCOMES:
Change in the health-related quality of life questionnaires of EQ-5D-5L in Chinese patients only | From Baseline to Week 33
  The change in the scores of the questionnaire EuroQol 5-Dimension 5-Level (EQ-5D-5L), including the health state index score (the higher, the better quality of life) and the visual anaglog scale (ranging from 0 to 100; the higher, the better quality of life).
Change in the health-related quality of life questionnaires of KDQoL-36 in Chinese only | From Baseline to Week 33
  The change in the scores of the questionnaire Kidney Disease Quality of Life 36-item short form (KDQoL-36). The score ranges from 0 to 100 for five domains, with higher scores indicating better quality of life.

CONTACTS AND LOCATIONS:
Locations (41):
- United States (18):
  - Renal Consultants Medical Group, Granada Hills, California
  - North America Research Institute - San Dimas, San Dimas, California
  - Rocky Mountain Kidney Care - Lone Tree, Lone Tree, Colorado
  - PACT Kidney Care - Orange, Orange, Connecticut
  - US Renal Care - Fort Myers South, Fort Myers, Florida
  - Nephrology & Hypertension Specialists, Dalton, Georgia
  - Renal Associates Of Baton Rouge, LLC, Baton Rouge, Louisiana
  - Nephrology Associates, P.C. - Columbus, Columbus, Mississippi
  - Nephrology & Hypertension Associates Ltd - Tupelo, Tupelo, Mississippi
  - High Desert Nephrology Association - US Renal Care, Gallup, New Mexico
  - US Renal Care - West Cheektowaga, Cheektowaga, New York
  - NY Kidney & Hypertension Medicine, Ridgewood, New York
  - US Renal Care - Alexis, Toledo, Ohio
  - Dallas Renal Group - Dallas, Dallas, Texas
  - US Renal Care - Bluebonnet, Fort Worth, Texas
  - Gamma Medical Research, McAllen, Texas
  - US Renal Care - South San Antonio, San Antonio, Texas
  - US Renal Care - Hill Country, San Antonio, Texas
- China (23):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Beijing Tsinghua Chang Gung Hospital, Beijing, Beijing Municipality
  - Peking University International Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Zhengzhou University-First Affiliated Hospital, Zhengzhou, Henan
  - Huazhong University of Science and Technology-Tongji Medical College - Wuhan Union Hospital, Wuhan, Hubei
  - Wuhan University People's Hospital, Wuhan, Hubei
  - Central South University-The Third Xiangya Hospital, Changsha, Hunan
  - Southeast University-Zhongda Hospital, Nanjing, Jiangsu
  - Jiangsu Province Hospital (The First Affiliated Hospital with Nanjing Medical University), Nanjing, Jiangsu
  - Nantong University-Affiliated Hospital, Nantong, Jiangsu
  - Nanjing Medical University-Wuxi People's Hospital (Wuxi No.1 People's Hospital), Wuxi, Jiangsu
  - Subei People's Hospital, Yangzhou, Jiangsu
  - Jiangxi Provincial People's Hospital, Nanchang, Jiangxi
  - Qingdao University-The Affiliated Hospital, Qingdao, Shandong
  - Yantai Yuhuangding Hospital, Yantai, Shandong
  - Shanghai Jiao Tong University School of Medicine (SJTUSM)-Renji Hospital, Shanghai, Shanghai Municipality
  - Fudan University-Zhongshan Hospital, Shanghai, Shanghai Municipality
  - Fudan University-Huashan Hospital, Shanghai, Shanghai Municipality
  - Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Tongren Hospital, Shanghai, Shanghai Municipality
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan